CLINICAL TRIAL: NCT05207436
Title: Pilot Test of Intranasal Oxytocin as an Enhancer of Brief Couples Therapy for PTSD
Brief Title: Brief Cognitive Behavioral Conjoint Therapy for PTSD With Adjunctive Intranasal Oxytocin
Acronym: CBCT+OT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Leslie Morland, Director of Telemental Health, Staff Clinical Psychologist, San Diego Veterans Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1227284
Record Dates: First submitted 2022-01-06; First posted 2022-01-26 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Post Traumatic Stress Disorder; Relational Problems
Keywords: Post Traumatic Stress Disorder; Oxytocin; Marital Therapy; Couples; Veterans; Telemedicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brief Cognitive Behavioral Conjoint Therapy for PTSD plus Intranasal Oxytocin (Experimental): Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (B-CBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Brief Cognitive-Behavioral Conjoint Therapy

INTERVENTIONS:
Drug: Oxytocin nasal spray — Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each B-CBCT session.
  Other Names: Pitocin
Behavioral: Brief Cognitive-Behavioral Conjoint Therapy — Eight sessions of standardized B-CBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
  Other Names: B-CBCT

SUMMARY:
In 2019 VA mandated that all Veterans seeking mental health care have access to flexible family mental health services in VA (VHA directive 1163.04). This study aims to respond to this mandate by further improving an evidence-based PTSD treatment designed to decrease PTSD symptoms and improve relationship satisfaction for Veterans and their romantic partners. Brief Cognitive-Behavioral Conjoint Therapy (B-CBCT), an 8-session dyadic psychotherapy for PTSD, has been found to significantly reduce PTSD symptoms, but the effects of B-CBCT on relationship satisfaction are less reliable and robust. Pharmacological augmentation of psychotherapy utilizing intranasal oxytocin, a neurohormone that influences mechanisms of trauma recovery and social behavior, may help improve relationship satisfaction outcomes. If successful, the proposed study will advance knowledge of strategies for improving Veterans' quality of life by improving their intimate relationships along with PTSD symptoms.

DETAILED DESCRIPTION:
Military Veterans often experience challenges reintegrating into their communities after military service, due in part to mental health problems such as posttraumatic stress disorder (PTSD). PTSD, a psychiatric disorder that develops in response to exposure to traumatic events, disproportionately affects Veterans, leads to poorer physical health, and impairs psychosocial functioning and quality of life. Mitigating the negative effects of PTSD on Veterans' health, functioning, and well-being is therefore a major goal of the VA.

The premise that interpersonal relationships play a key role in resilience, risk, and recovery from trauma is supported by research showing a robust association between PTSD and social support. Treatment approaches that bolster Veterans' internal strengths and enhance the capacity of their social environments to provide support are most likely to have powerful effects on well-being.

Many Service Members and Veterans with PTSD experience impairment and distress within intimate relationships at greater levels than among civilian couples. Consistent with this, Veterans seeking treatment for PTSD often identify relationships as targets of intervention and express the desire to involve close others in treatment. The VA has been responsive to these needs, as shown by the continuum of services available to Veterans and their families through the VA Family Services program. The Veterans' Mental Health and Other Care Improvements Act of 2008 stated that marriage and family counseling were to be available to Veterans to facilitate their treatment and rehabilitation. In 2009, VA began an initiative to select evidence-based family therapies and train mental health providers in these treatments. More recently, Directive 1163.04 indicated that Veterans with a mental health diagnosis should be asked about their interest in having family involved in their care and be offered marital and family counseling. The VA Family Services program supports several treatment approaches to meet the diverse mental health needs of Veterans and their loved ones. One such option for Veterans who want to simultaneously improve their PTSD symptoms and their relationship functioning is Cognitive-Behavioral Conjoint Therapy (CBCT) for PTSD. The VA has been disseminating CBCT since 2013.

CBCT is a PTSD-specific cognitive-behavioral psychotherapy attended by the couple that uses close relationships as the vehicle for recovery. Across 15 75-minute sessions, this manualized therapy addresses the patient's PTSD and relationship functioning simultaneously via its focus on PTSD psychoeducation within relationship contexts, communication skills, behavioral approach exercises, and cognitive interventions. CBCT effectively treats PTSD, exhibiting large within-group effect sizes on clinician-rated PTSD symptoms.

Across studies, however, CBCT has had less robust, more variable effects on relationship satisfaction than on PTSD. This is likely because the factors governing relationship satisfaction are complex and rely on a number of independent, interpersonal factors. The largest published study of CBCT (N = 40 dyads), in which CBCT was compared to a waitlist control group, found a moderate within-group effect (g = 0.64) and between-group effect (g = 0.47) of CBCT on Veterans' relationship satisfaction. This sample, however, was composed of only about 25% Veterans. Given that Veteran couples are known to have lower relationship satisfaction than non-Veteran couples, it is important to further examine CBCT among Veteran couples that are more representative of couples seen in general VA practice to increase generalizability of findings. However, preliminary data from couples treated as part of VA's dissemination of CBCT suggest that effects on relationship satisfaction are noticeably smaller than in previous studies. This may be due, in part, to poor engagement in the intervention. Couples experience many logistical obstacles to engaging in care (e.g., the need to coordinate schedules, lack of childcare). Veterans with PTSD can encounter additional obstacles related to beliefs about mental health and mental health treatment.

To address these obstacles to treatment engagement, Dr. Leslie Morland (PI) recently completed a study of an 8-session version of CBCT (B-CBCT) delivered either in-office or via telehealth to home compared to a family education control condition. She and her team similarly found robust reductions in PTSD symptoms in B-CBCT (B-CBCT within-group d's = 1.05-1.12, between-group d's = 0.59-0.76) but only a small effect on both partners' relationship satisfaction that was on par with the family education condition (B-CBCT within-group d = 0.38; between-group d's = 0.04-0.12).

Medications that potentiate the mechanisms of action in psychotherapy could enhance their effects. The neuropeptide oxytocin appears to be a promising medication because it mediates processes central to PTSD and relationship functioning. Oxytocin is a 9-amino-acid nonapeptide hormone produced by the paraventricular and supraoptic nuclei of the hypothalamus that regulates human emotions, social cognition, and social behaviors. Endogenous oxytocin assists in milk production for breastfeeding, induces contractions during childbirth, is released during orgasm, may reduce urine volume, and may induce sodium release from the kidneys. Intravenous oxytocin is used in medical practice to induce labor in pregnant women and to increase muscle tone in the uterus in the case of postpartum bleeding. Oxytocin is released to several brain areas, including the amygdala, hypothalamus, hippocampus, insula, and striatum, and effects are mediated by oxytocin receptors found in these regions.

Intranasal administration of oxytocin may offer understanding of the causal effects of oxytocin on human behavior. Intranasal oxytocin is safe and easy to administer, with a short half-life that makes it highly suitable for adding to behavioral interventions. Intranasal oxytocin is best known for its widespread effects on affiliative processes and behaviors. For example, intranasal oxytocin increases trust, empathy, generosity, positive communication, and emotional disclosure. Oxytocin also improves social cognition, including emotion recognition and empathic accuracy. The combination of intranasal oxytocin with provision of social support suppresses cortisol release and subjective responses to social stress.

Intranasal oxytocin can be conceptualized as a "psychotherapy process catalyst", in that oxytocin could enhance patients' openness to intervention, attention to others' communication, and willingness and ability to develop therapeutic alliance. A recent systematic review of 14 studies of the effects of intranasal oxytocin on PTSD symptoms concluded that there is tentative evidence for the clinical utility of intranasal oxytocin for PTSD, although more studies with chronic administration are needed. To date, only one pilot study has examined the effects of oxytocin-enhanced psychotherapy for PTSD. Findings indicated that participants randomized to Prolonged Exposure (PE) for PTSD augmented with oxytocin demonstrated lower PTSD and depression symptoms and had higher working alliance scores compared to participants randomized to PE with placebo. A large, two-site phase II randomized controlled trial (RCT) of oxytocin-enhanced PE is currently being conducted in the VA by a Collaborator on this project (PI: Dr. Julianne Flanagan; NCT04228289).

Administering intranasal oxytocin in a safe, therapeutic context in which interpersonal skill-building takes place is hypothesized to lead to prosocial effects and facilitated recovery. CBCT is therefore the ideal treatment platform for oxytocin augmentation. CBCT and oxytocin are both inherently interpersonal and could operate in a coordinated, synergistic manner to improve relationship satisfaction. For example, facilitating positive communication could enhance all aspects of the therapy, including both partners' sharing of thoughts and feelings and their ability to join together in cognitive restructuring of trauma-related beliefs that interfere with recovery. Findings that intranasal oxytocin increases neural activation to socially rewarding stimuli and facilitates social approach behavior suggest that it could help Veterans and their partners embrace social situations, which is central to CBCT behavioral interventions. Lastly, generalization of improvements in trust, empathy, positive communication, and approach behavior could help Veterans participate more fully with their families (e.g., improved parenting skills) and many other domains of society (e.g., education and employment). To date, however, oxytocin has not been tested as an adjuvant to CBCT nor any relationship-focused therapy for trauma-exposed Veterans.

Based on compelling pre-clinical data implicating the oxytocin system in affiliative behavior, the study of intranasal oxytocin in humans expanded very rapidly. However, these developments were followed by calls for caution after acknowledgment of lack of replicability of findings, methodological limitations such as low statistical power, and poor understanding of the pharmacodynamics of intranasal delivery of synthetic oxytocin. Intranasal oxytocin is thought to exert effects by bypassing the blood-brain barrier and reaching the brain directly (i.e., nose-to-brain transport), but definitive data have been lacking. More recently, pre-clinical, primate, and human research have converged to indicate that intranasal oxytocin does, in fact, reach the brain to a degree that leads to clinically relevant changes in behavior, ostensibly through olfactory and trigeminal nerve fibers. Another issue that has affected the translation of oxytocin research to treatment has been the lack of dose-ranging studies in humans. Notably, most intranasal oxytocin studies have administered only one dose of intranasal oxytocin, typically 24 or 40 international units. The pharmacodynamics of repeated oxytocin administration are not well-established, but given the short half-life of intranasal oxytocin (i.e., 20 or more minutes in cerebrospinal fluid and 2 minutes in blood), repeated dosing (e.g., daily, weekly) is not hypothesized to operate differently than single doses.

The proposed study to augment CBCT with intranasal oxytocin and to examine its effects on intimate relationship adjustment, social functioning more generally, and quality of life directly addresses the mission of the VA, as outlined in the VA fiscal year (FY) 2018-2024 Strategic Plan. Specifically, the proposed study seeks to advance knowledge of how to help Veterans have good quality of life-which the VA identifies as including satisfying relationships-in three ways: First, findings will inform whether B-CBCT social functioning outcomes can be improved with adjunctive medication. Second, if oxytocin enhances the mechanisms described in this proposal as predicted, it could further strengthen rationale for providers administering eight-session B-CBCT rather than 15-session CBCT. Effectively truncating CBCT would mean that more patients could be seen by the same number of VA providers, potentially improving Veterans' access to treatment. Greater effectiveness and efficiency of treatment could lead to lower costs to VA. Third, by targeting mechanisms that are salient to all interpersonal relationships (e.g., trust), oxytocin could help the effects of CBCT extend to non-intimate relationships, thereby improving overall quality of life and potentially having effects on other issues facing the VA (such as suicide) which is known to be related to interpersonal difficulties. Lastly, improving Veterans' social environments could help them maintain their gains and respond effectively to future stressors-potentially lowering the likelihood of future need for episodes of care.

ELIGIBILITY:
Inclusion Criteria:

* One member of the couple be a Veteran enrolled in the San Diego VA Healthcare System with a Posttraumatic Stress Disorder Checklist-5 score of > 33, indicating a likely PTSD diagnosis.
* Agree not to receive other individual or conjoint psychotherapy for PTSD during the treatment portion of the study
* If already on psychoactive medication prior to study referral, Veteran participant must remain on a stable psychoactive medication regimen for at least 45 days.

Exclusion Criteria:

* Acute suicidality
* Psychosis
* Active substance use disorder
* Severe ongoing medical problems, including heart disease and neuroendocrinological disorders (e.g., diabetes)
* Uncontrolled hypotension (systolic blood pressure <100 mm Hg) or hypertension (>160/100 mm Hg)
* Pregnancy, delivery in the past 6 months, or current breastfeeding
* Severe intimate aggression reported by either partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morland, PsyD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brief Cognitive Behavioral Conjoint Therapy for PTSD Plus Intranasal Oxytocin
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 10 couples (20 individuals)
Arm/Group | Brief Cognitive Behavioral Conjoint Therapy for PTSD Plus Intranasal Oxytocin
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.10 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Couples Satisfaction Inventory-32
Description: The Couples Satisfaction Index is a 32-item self-report survey assessing several domains of relationship satisfaction. Higher sum scores (range 0 to 161) represent higher relationship satisfaction.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- bCBCT+OT-Veterans; bCBCT+OT-Partners: Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Oxytocin (OT) nasal spray: Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each bCBCT session.
  Brief Cognitive-Behavioral Conjoint Therapy: Eight sessions of standardized bCBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 103.6 (32.17) | 87.30 (36.70)

2. Primary Outcome: Couples Satisfaction Inventory-32
Description: as for outcome 1
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 124.67 (23.70) | 113.44 (39.08)

3. Primary Outcome: Couples Satisfaction Inventory-32
Description: as for outcome 1
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 114.38 (40.90) | 113.0 (49.50)

4. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (PCL-5)
Description: The PCL-5 is a 20-item self-report questionnaire assessing symptoms of PTSD based on DSM-V criteria. Scores range from 0 to 80, with higher scores representing more severe symptoms.
Time Frame: baseline
Population: Veteran data only; partner PCL-5 not an outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans
Number analyzed (Participants) | 10
score on a scale | 47.78 (10.12)

5. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 4
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Population: Veterans only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans
Number analyzed (Participants) | 10
score on a scale | 25.44 (13.23)

6. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: as for outcome 4
Time Frame: three months post-treatment (approximately 5-months after baseline)
Population: Veterans only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans
Number analyzed (Participants) | 10
score on a scale | 31.22 (14.94)

7. Secondary Outcome: Brief Inventory of Psychosocial Functioning
Description: The Brief Inventory of Psychosocial Functioning (B-IPF) is a 7-item self-report measure designed to assess multiple dimensions of functional impairment related to psychiatric disturbances. Higher scores (range 0 to 100) indicate more functional impairment.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- bCBCT-OT-Veterans; bCBCT+OT-Partners: Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Oxytocin (OT) nasal spray: Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each bCBCT session.
  Brief Cognitive-Behavioral Conjoint Therapy: Eight sessions of standardized bCBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
Arm/Group | bCBCT-OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 50.49 (20.03) | 31.22 (21.25)

8. Secondary Outcome: Brief Inventory of Psychosocial Functioning
Description: as for outcome 7
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 31.58 (27.35) | 20.37 (14.87)

9. Secondary Outcome: Brief Inventory of Psychosocial Functioning
Description: as for outcome 7
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- bCBCT+OT--Partners: Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (bCBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Oxytocin (OT) nasal spray: Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each bCBCT session.
  Brief Cognitive-Behavioral Conjoint Therapy: Eight sessions of standardized bCBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT--Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 32.00 (27.39) | 23.81 (23.15)

10. Other Pre Specified Outcome: World Health Organization Quality of Life - Brief (BREF) - Physical
Description: The World Health Organization Quality of Life - BREF - Physical is a 7-item self-report questionnaire assessing an individual's physical health and functioning. Scores range from 0 to 100, with higher scores representing a better outcome
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 50.19 (9.28) | 42.21 (9.91)

11. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Physical
Description: as for outcome 10
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 55.16 (6.94) | 55.56 (11.02)

12. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Physical
Description: as for outcome 10
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT--Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 51.98 (10.58) | 54.02 (9.04)

13. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Psychological
Description: The World Health Organization Quality of Life - BREF - Psychological is a 6-item self-report questionnaire that assesses an individual's mental well-being and psychological functioning. Scores range from 0 to 100, with higher scores representing a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 51.39 (11.41) | 62.04 (14.20)

14. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Psychological
Description: as for outcome 13
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 54.17 (12.67) | 65.74 (17.02)

15. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Psychological
Description: as for outcome 13
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT--Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 52.78 (13.98) | 65.10 (10.67)

16. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Social
Description: The World Health Organization Quality of Life - BREF - Social is a 3-item self-report questionnaire that assesses an individual's satisfaction with their social relationships. Scores range from 0 to 100, with higher score representing a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 47.92 (20.77) | 50.00 (23.57)

17. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Social
Description: as for outcome 16
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 65.63 (20.14) | 62.04 (27.67)

18. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Social
Description: as for outcome 16
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 57.41 (18.84) | 66.67 (23.15)

19. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Environment
Description: The World Health Organization Quality of Life - BREF - Environmental is an 8-item self-report questionnaire that assesses an individual's satisfaction with their physical, social, and home environment. Scores range from 0 to 100, with higher scores representing a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 65.28 (11.63) | 68.06 (17.59)

20. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Environment
Description: as for outcome 19
Time Frame: immediately after the intervention (approximately 2-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 72.22 (11.42) | 72.92 (16.83)

21. Other Pre Specified Outcome: World Health Organization Quality of Life - BREF - Environment
Description: as for outcome 19
Time Frame: three months post-treatment (approximately 5-months after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBCT+OT-Veterans | bCBCT+OT-Partners
Number analyzed (Participants) | 10 | 10
score on a scale | 64.93 (18.74) | 72.66 (14.44)

ADVERSE EVENTS:
Time Frame: 11 weeks
Groups:
- bCBCT-OT-Veteran: Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (B-CBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Oxytocin nasal spray: Veteran participants will self-administer 40 IU of intranasal oxytocin 30 minutes before the start of each B-CBCT session.
  Brief Cognitive-Behavioral Conjoint Therapy: Eight sessions of standardized B-CBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
- bCBCT-OT-Partner: Couples will receive Brief Cognitive-Behavioral Conjoint Therapy (B-CBCT) weekly. Prior to each session, the Veteran participant will self-administer intranasal oxytocin. The estimated length of treatment participation is 8 to 15 weeks. All procedures take place in the Veterans home via home-based clinical video teleconferencing (CVT).
  Oxytocin nasal spray: Veteran participants only.
  Brief Cognitive-Behavioral Conjoint Therapy: Eight sessions of standardized B-CBCT, a manualized couple-based intervention for PTSD designed to simultaneously reduce PTSD and enhance relationship and functioning.
Arm/Group | bCBCT-OT-Veteran | bCBCT-OT-Partner
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | bCBCT-OT-Veteran (N=10) | bCBCT-OT-Partner (N=10)
pounding heart (Cardiac disorders) | 1 (1) | NA — one veteran sought medical attention for a "pounding heart" after session 4 of bCBCT+OT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05207436/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT05207436/SAP_001.pdf